CLINICAL TRIAL: NCT01491997
Title: Mind-Body Medicine and Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Ali Keshavarzian, Director, Division of Digestive Diseases, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AT11-003 - 1 R01 AT007143-01
Record Dates: First submitted 2011-12-07; First posted 2011-12-14 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mind Body Medicine Course 1 (Active Comparator): The subject of each course is Mind/Body medicine. One course is learning about the mind and the body through experiences. The other is learning about the mind and the body through experiences. Both courses will follow the same format, meeting once every week, for a total of 8 weeks, for roughly 2 hours per class. You will be provided with a schedule of the weekly classes, which will occur on the same day every week, at the same time. Weekly sessions will be run by a teacher and will include other participants in the class. . You will also be given homework assignments that are intended to reinforce what you learn in the program. The assignments will require up to 45 minutes, 6 days/week. Following the 6th class, and before the 7th class, there is a voluntary ½ day Saturday program. Participation in this program is optional. You are expected to continue to incorporate what you learned in the class in your daily routine after you are done with the classes.
  Interventions: Behavioral: Mind/Body Medicine Course 1
- Mind/Body Medicine Course 2 (Active Comparator): The subject of the course is Mind/Body medicine. This course is learning about the mind and the body through lectures. The course will meet once every week, for a total of 8 weeks, for roughly 2 hours per class. You will be provided with a schedule of the weekly classes, which will occur on the same day every week, at the same time. Weekly sessions will be run by a teacher and will include other participants in the class. You will also be given homework assignments that are intended to reinforce what you learn in the program. The assignments will require up to 45 minutes, 6 days/week. Following the 6th class, and before the 7th class, there is a voluntary all day Saturday program. Participation in this program is optional. You are expected to continue to incorporate what you learned in the class in your daily routine after you are done with the classes.
  Interventions: Behavioral: Mind/Body Medicine Course 2

INTERVENTIONS:
Behavioral: Mind/Body Medicine Course 1 — The subject of the course is Mind/Body medicine. This course is learning about the mind and the body through experiences. The course will meet once every week, for a total of 8 weeks, for roughly 2 hours per class. You will be provided with a schedule of the weekly classes, which will occur on the same day every week, at the same time. Weekly sessions will be run by a teacher and will include other participants in the class. You will also be given homework assignments that are intended to reinforce what you learn in the program. The assignments will require up to 45 minutes, 6 days/week. Following the 6th class, and before the 7th class, there is a voluntary all day Saturday program. Participation in this program is optional. You are expected to continue to incorporate what you learned in the class in your daily routine after you are done with the classes.
  Arms: Mind Body Medicine Course 1
Behavioral: Mind/Body Medicine Course 2 — The subject of the course is Mind/Body medicine. This course is learning about the mind and the body through lectures. The course will meet once every week, for a total of 8 weeks, for roughly 2 hours per class. You will be provided with a schedule of the weekly classes, which will occur on the same day every week, at the same time. Weekly sessions will be run by a teacher and will include other participants in the class. You will also be given homework assignments that are intended to reinforce what you learn in the program. The assignments will require up to 45 minutes, 6 days/week. Following the 6th class, and before the 7th class, there is a voluntary all day Saturday program. Participation in this program is optional. You are expected to continue to incorporate what you learned in the class in your daily routine after you are done with the classes.
  Arms: Mind/Body Medicine Course 2

SUMMARY:
Stress has been linked to chronic health problems, particularly diseases involving inflammation-mediated tissue injury and organ failure. Accordingly, it is not surprising that mind/body interventions are advocated for treatment of chronic inflammatory diseases. One such candidate disease is ulcerative colitis (UC) because: (1) UC is a life-long, relapsing, disabling inflammatory disorder of the intestine that lacks a non-toxic, efficacious treatment; (2) the therapeutic goal is to improve quality of life by ameliorating disabling symptoms and preventing disease progression by preventing disease flare-up, (3) stress triggers UC flare-up by modifying intestinal function and inflammatory processes, highlighting the potential therapeutic benefit of reducing physiological stress responses. The purpose of this study is to see if either of two 8-week mind/body medicine courses has an effect in reducing stress and affecting the course and severity of UC. Both have been shown to benefit other aspects of health and well-being.

DETAILED DESCRIPTION:
Statistical Analysis. The investigator will use the biopsychomarkers identified as the highest prediction value to determine the relative accuracy to predict response to the Mindful Intervention (i.e., disease outcome). For response to the mindful intervention, the investigator will use the use the combination of markers to study whether they correctly predict the response to the intervention. The investigator will study the accuracy of the markers using area under the curve (AUC) summary index for ROC curves.181 If the classification accuracy of the markers is high then the area under the curve will be close to 1. If the predictive accuracy of the combined set of markers were poor then the (AUC) will be close to 0.5.

Power Estimates UC disease flare-up was quite common in this sample, occurring in well over half of subjects in the samples collected in the discovery phase. The power analyses, assuming α = 0.05 for all tests indicated that for models involving analyses of correlational data, there will be sufficient power at even small effect sizes for the smallest possible sample with full data across all data points and virtually all variables. For the most conservative estimate, the investigator base their calculations on having 50 participants with data with full integrity. With an effect size of r = 0.15 and n = 50, power is 80 or greater to detect effect sizes of r = 0.20. Effect sizes below this threshold would likely not be clinically significant or substantively interpretable, as they would explain less than 2% in the variance of the dependent variable. Thus, most effect sizes that would be reasonably and substantially interpretable will have good power. Each factor that is suspected of varying between groups can be examined with the chi-square test based on 1 degrees of freedom, by setting it invariant in one model and then allowing it to be freely estimated in the other. Such a chi-square test provides a power of 0.80 with effect size difference of 0.15.

For binary categorical measures, such as responsiveness to MSRB, the investigator conducted separate power analyses.

The power for adjusted analyses of primary predictors of interest will be evaluated as a function of the risk of outcome when all ancillary variables are set to their mean value, the predictor is set to the mean value, and proportion of variance in predictor explained by the ancillary variables, and the odds ratio of outcome variable from increasing the predictor by an amount equal to one of its standard deviation. The range in probabilities of outcome variables can be anywhere from 20% for less likely events and 50% for more likely events, the investigator will provide power calculations over a wide range of probabilities. The investigator believe that the amount of variation of our typical model ranges from about 20% to 50%. The table (below) represents the minimum odds ratio than can be detected with 80% power, which indicate good power for expected outcome.

Proportions R2 =.20 R2=.50 0.10 1.64 1.87 0.20 1.46 1.63 0.30 1.39 1.53 0.40 1.35 1.48 0.50 1.32 1.43

ELIGIBILITY:
Inclusion Criteria:

* You have been diagnosed with moderately severe Ulcerative Colitis at the time of your last flare up
* You experienced at least one flare-up within the last year
* Either no IBD medication or have been on a stable dose of oral 5-ASA products (i.e. Mesalamine, Sulfasalazine, or Colazol) for at least 3 weeks, immunomodulators (Imuran, 6MP, Methotrexate)for at least 3 months and biologics (TNF antibody) for at least 6 months prior to enrollment
* If on maintenance 5-ASA products or immunomodulators and dose changes during the study, participant agrees to remain on that dose for the study duration
* ACTIVE UC PATIENTS: If on Prednisone the dose must not be more than 20mg/day; you can be weaned off Prednisone by 5mg/day weekly to 10mg/day weekly to 2.5mg/day weekly

Exclusion Criteria:

* Other forms of colitis, such as Clostridium Difficile Colitis or Indeterminate Colitis
* Current use of oral steroids within the last 30 days, topical agents (i.e. steroids or 5-ASA) within the last 14 days
* History of colon resection
* Antibiotic use within the last 14 days
* WOMEN: Cannot be pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Biopsychomarkers | 4 years
  Develop a set of biopsychomarkers to (a) identify characteristics that predict UC patient's response to Mind/Body Medicine courses and (b) establish an objective set of markers that demonstrate the impact of Mind/Body Medicine courses on well-being and UC disease state.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Keshavarzian, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Jedel S, Beck T, Swanson G, Hood MM, Voigt RM, Gorenz A, Jakate S, Raeisi S, Hobfoll S, Keshavarzian A. Mindfulness Intervention Decreases Frequency and Severity of Flares in Inactive Ulcerative Colitis Patients: Results of a Phase II, Randomized, Placebo-Controlled Trial. Inflamm Bowel Dis. 2022 Dec 1;28(12):1872-1892. doi: 10.1093/ibd/izac036. PMID 35661212